CLINICAL TRIAL: NCT06754280
Title: Developing a Sedentary Reducing Intervention for Black Adults With CKD: RESET-CKD
Brief Title: An Intervention to Reduce Sedentary Behavior for Black Adults With Chronic Kidney Disease
Acronym: RESET-CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Mary Hannan, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-1410; K23NR021034 (NIH)
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease(CKD)
Keywords: Sedentary
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RESET-CKD (Experimental): RESET-CKD is a 12-week intervention that consists of four major components to support decreasing sedentary behavior: (1) health coaching, (2) feedback charts on sedentary behavior, (3) a workbook, and (4) reminders and cues.
  Interventions: Behavioral: RESET-CKD
- Attention Control (Active Comparator): CKD-related education
  Interventions: Other: Attention Control

INTERVENTIONS:
Behavioral: RESET-CKD — RESET-CKD is a 12-week intervention that consists of four major components to support decreasing sedentary behavior: (1) health coaching, (2) feedback charts on sedentary behavior, (3) a workbook, and (4) reminders and cues.
  Arms: RESET-CKD
Other: Attention Control — CKD-related education
  Arms: Attention Control

SUMMARY:
RESET-CKD is evaluating an intervention to support Black adults with chronic kidney disease (CKD) to reduce their sedentary (e.g., sitting) time. Half of the participants will be randomized to the intervention, where the goal is to support individuals to reduce their sitting time, and the other half will be randomized to an attention control condition that provides CKD-related education not related to sedentary behavior. All participants will be followed for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as Black or African American
* Age ≥35 to ≤80 years old
* CKD Stage 1-4
* Self-reported 6 or more hours/day of sedentary time
* Ability to speak/read/understand English
* Has access to a telephone

Exclusion Criteria:

* Being unable to walk 1 block
* Being unable to stand from a seated position without assistance
* Using a wheelchair, walker, or cane for all of their ambulation
* Presence of a condition(s) or diagnosis, either physical or psychological, that precludes participation, including: Lower-extremity amputation (AKA or BKA) without prosthetic, Orthopedic condition that would preclude prompted sit-to-stand transitions or standing, Neurologic or psychiatric condition that would preclude prompted sit-to- stand transitions or standing, Severe cognitive impairment, Unstable coronary artery disease (i.e., angina with activity), Orthostatic hypotension
* Kidney transplant
* Any other condition that the investigator considers precludes participation in the trial
* Participated in the Patient Advisory Board

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in sedentary time | Baseline to week 12
  Change in activPAL-measured sedentary time

SECONDARY OUTCOMES:
Change in self-reported sedentary time | Baseline to week 12
  Change in self-reported sedentary time
Change in health-related quality of life | Baseline to week 12
  Change in health-related quality of life measured via the KDQOL

CONTACTS AND LOCATIONS:
Locations (1):
- UI Health/University of Illinois Chicago, Chicago, Illinois, United States